CLINICAL TRIAL: NCT00759473
Title: D-Cycloserine Facilitation of Cocaine - Cue Extinction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Kathleen Brady, MD, PhD, Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HRs#17972, 19784; R01DA023188 (NIH)
Record Dates: First submitted 2008-09-24; First posted 2008-09-25 (Estimated); Results first posted 2013-07-10 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-03

CONDITIONS: Cocaine Use Disorders
Keywords: substance-related disorders
MeSH Terms: conditions — Substance-Related Disorders | interventions — Cycloserine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Placebo/Placebo/Placebo/Placebo (Placebo Comparator): Participants were assigned to receive placebo for each of 3 cue exposure sessions and at the one-week follow-up session. During cue exposure sessions, participants were asked to handle cocaine cues such as simulated crack, powder, and pipes while listening to an imagery script, and then they watched video footage of cocaine-related activities.
  Interventions: Drug: Placebo
- DCS/DCS/DCS/Placebo (Experimental): Participants were assigned to receive 50 mg of d-cycloserine (DCS) for each of 3 cue exposure sessions and a placebo at the one-week follow-up session. During cue exposure sessions, participants were asked to handle cocaine cues such as simulated crack, powder, and pipes while listening to an imagery script, and then they watched video footage of cocaine-related activities.
  Interventions: Drug: D-Cycloserine (DCS)
- DCS/Placebo/DCS/Placebo (Other): Participants were assigned to receive 50 mg of d-cycloserine (DCS) at the first and third cue exposure sessions and a placebo at the second cue exposure and the one-week follow-up session. During cue exposure sessions, participants were asked to handle cocaine cues such as simulated crack, powder, and pipes while listening to an imagery script, and then they watched video footage of cocaine-related activities.
  Interventions: Drug: D-Cycloserine (DCS)
- DCS/DCS/Placebo (Experimental): Participants were assigned to receive 50 mg of d-cycloserine (DCS) for each of 2 cue exposure sessions and a placebo at the one-week follow-up session. During cue exposure sessions, participants were asked to handle cocaine cues such as simulated crack, powder, and pipes while listening to an imagery script, and then they watched video footage of cocaine-related activities. Cue exposure sessions were accompanied by instructions on coping with craving.
  Interventions: Drug: D-Cycloserine (DCS)
- Placebo/Placebo/Placebo (Active Comparator): Participants were assigned to placebo for each of 2 cue exposure sessions and a placebo at the one-week follow-up session. During cue exposure sessions, participants were asked to handle cocaine cues such as simulated crack, powder, and pipes while listening to an imagery script, and then they watched video footage of cocaine-related activities. Cue exposure sessions were accompanied by instructions on coping with craving.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: D-Cycloserine (DCS) — 50 mg d-cycloserine or placebo taken orally
  Other Names: seromycin
  Arms: DCS/DCS/DCS/Placebo; DCS/DCS/Placebo; DCS/Placebo/DCS/Placebo
Drug: Placebo
  Arms: Placebo/Placebo/Placebo; Placebo/Placebo/Placebo/Placebo

SUMMARY:
The purpose of this study is to explore the use of d-cycloserine (DCS) to facilitate extinction of response to cocaine cues in cocaine-dependent individuals, in hopes that it may lead to the development of new treatment options for cocaine dependence.

DETAILED DESCRIPTION:
Cocaine dependence remains a serious problem in the United States today and in spite of two decades of intense research, efficacious pharmacotherapeutic treatments have not been identified. Cocaine-associated environmental cues can elicit drug craving and exposure to cocaine-related cues is likely to be involved in relapse. Emerging data supports the role of glutamate in extinction learning. D-cycloserine (DCS), a partial glutamate agonist, facilitates extinction of associative learning in animal models of fear-conditioning and clinical studies of exposure treatment for anxiety disorders. A recent study demonstrated DCS acceleration of extinction of cocaine-induced conditioned place preference in rats (Botreau et al., 2006). Exploration of DCS in facilitating extinction of response to drug-related cues in humans is needed. The proposed study will extend these innovative and promising findings from the basic science arena and anxiety disorders field in a proof of concept investigation of DCS facilitation of extinction of response to cocaine-related cues in a human laboratory paradigm. In addition, to examine the neural substrates of extinction learning, a sub-set of individuals that are willing and eligible will undergo fMRI scanning procedures before and after the extinction protocol.

ELIGIBILITY:
Inclusion Criteria

1. Subjects must be able to provide informed consent and function at an intellectual level sufficient to allow accurate completion of all assessment instruments.
2. Subjects must meet DSM-IV criteria for current cocaine dependence. Subjects may meet criteria for abuse, but not dependence on any other substance with the exceptions of nicotine and alcohol. Because of the high comorbidity of cocaine with alcohol and nicotine dependence, excluding nicotine and alcohol dependence would seriously compromise the feasibility of recruitment. Nicotine use immediately prior to the cue exposure/extinction session will be controlled. Although individuals who meet criteria for alcohol dependence will be accepted for study participation, anyone who has a measurable blood alcohol level on the day of the sessions will be excluded as acute alcohol intake can increase serum levels of DCS and lower the seizure threshold.
3. Use of one of the following methods of birth control by female subjects: birth control pills, barrier methods (diaphragm or condoms with spermicide or both), surgical sterilization, use of an intra-uterine contraceptive device, or complete abstinence from sexual intercourse.
4. Subjects must live within a 50-mile radius of the research facility and have reliable transportation.
5. Subjects must consent to remain abstinent from all drugs of abuse (except nicotine) prior to the first session and through the final session.
6. Subjects must consent to random assignment to the DCS vs. placebo conditions.
7. For fMRI participants, subjects must be right-handed.

Exclusion Criteria

1. Women who are pregnant, nursing or of childbearing potential and not practicing an effective means of birth control.
2. Subjects with evidence of or a history of significant hematological, endocrine, cardiovascular, pulmonary, renal, gastrointestinal, or neurological disease including insulin-dependent diabetes, as these conditions may affect heart rate or skin conductance measurement.
3. Subjects with a history of or current psychotic disorder, current major depressive disorder, bipolar affective disorder or a severe anxiety disorder as these may impact cue reactivity.
4. Subjects who are unwilling or unable to maintain abstinence from alcohol and other drugs of abuse (except nicotine) prior to and between the cue procedures.
5. Subjects meeting DSM-IV criteria for substance dependence (other than nicotine, alcohol or cocaine as appropriate) within the past 60 days.
6. Subjects currently taking B-blockers, anti-arrhythmic agents, psychostimulants or any other agents known to interfere with heart rate and skin conductance monitoring.
7. Known or suspected hypersensitivity to DCS.
8. Individuals taking medications that could adversely interact with study medications, including, but not limited to ethionamide, isoniazid, or amino acid supplements.
9. Subjects with a history of epilepsy or seizure disorder.
10. Subjects with significant liver impairment, as DCS may increase serum transaminases.
11. For fMRI participants, the need for maintenance or acute treatment with any psychoactive medication including anti-seizure medications which could potentially interfere with fMRI.
12. For fMRI participants, clinically significant psychiatric or medical problems that would impair participation or limit ability to participate in scan.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2008-09; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen T Brady, M.D., Ph.D., Principal Investigator — Medical University of South Carolina
Locations (2):
- United States (2):
  - Medical University of South Carolina, Charleston, South Carolina
  - Behavioral Health Services of Pickens County, Pickens, South Carolina

REFERENCES:
- [Derived] Prisciandaro JJ, Joseph JE, Myrick H, McRae-Clark AL, Henderson S, Pfeifer J, Brady KT. The relationship between years of cocaine use and brain activation to cocaine and response inhibition cues. Addiction. 2014 Dec;109(12):2062-70. doi: 10.1111/add.12666. Epub 2014 Jul 21. PMID 24938849
- [Derived] Prisciandaro JJ, Myrick H, Henderson S, McRae-Clark AL, Santa Ana EJ, Saladin ME, Brady KT. Impact of DCS-facilitated cue exposure therapy on brain activation to cocaine cues in cocaine dependence. Drug Alcohol Depend. 2013 Sep 1;132(1-2):195-201. doi: 10.1016/j.drugalcdep.2013.02.009. Epub 2013 Mar 14. PMID 23497788

RESULTS

PARTICIPANT FLOW:
Groups:
- DCS/DCS/DCS/ Placebo: Participants were assigned to receive 50 mg of d-cycloserine (DCS) for each of 3 cue exposure sessions and a placebo at the one-week follow-up session. During cue exposure sessions, participants were asked to handle cocaine cues such as simulated crack, powder, and pipes while listening to an imagery script, and then they watched video footage of cocaine-related activities.
- Placebo/Placebo/Placebo/Placebo: Participants were assigned to receive a placebo for each of 3 cue exposure sessions and at the one-week follow-up session.During cue exposure sessions, participants were asked to handle cocaine cues such as simulated crack, powder, and pipes while listening to an imagery script, and then they watched video footage of cocaine-related activities.
- DCS/ Placebo/DCS/Placebo: Participants were assigned to receive 50 mg of d-cycloserine (DCS) at the 1st and 3rd cue sessions and placebo at the 2nd cue session and the one-week follow-up session. During cue exposure sessions, participants were asked to handle cocaine cues such as simulated crack, powder, and pipes while listening to an imagery script, and then they watched video footage of cocaine-related activities.
- DCS/DCS/Placebo: Participants were assigned to receive 50 mg of d-cycloserine (DCS) at 2 cue cue exposure sessions, and placebo at the one-week follow-up session. During cue exposure sessions, participants were asked to handle cocaine cues such as simulated crack, powder, and pipes while listening to an imagery script, and then they watched video footage of cocaine-related activities. Cue exposure was accompanied by instructions on how to cope with craving.
- Placebo/Placebo/Placebo: Participants were assigned to receive placebo at 2 cue exposure sessions, and at the one-week follow-up session. Participants also received cognitive skills training. During cue exposure sessions, participants were asked to handle cocaine cues such as simulated crack, powder, and pipes while listening to an imagery script, and then they watched video footage of cocaine-related activities. Cue exposure was accompanied by instructions on how to cope with craving.
Period: Overall Study
Arm/Group | DCS/DCS/DCS/ Placebo | Placebo/Placebo/Placebo/Placebo | DCS/ Placebo/DCS/Placebo | DCS/DCS/Placebo | Placebo/Placebo/Placebo
Started | 10 | 10 | 12 | 23 | 24
Completed | 10 | 10 | 12 | 23 | 24
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- DCS/DCS/DCS/Placebo: Participants were assigned to receive 50 mg of DCS for each of 3 cue exposure sessions and a placebo at the one-week follow-up session.During cue exposure sessions, participants were asked to handle cocaine cues such as simulated crack, powder, and pipes while listening to an imagery script, and then they watched video footage of cocaine-related activities.
- DCS/ Placebo/DCS/Placebo: Participants were assigned to receive 50 mg of DCS at the 1st and 3rd cue sessions and placebo at the 2nd cue session and the one-week follow-up session.During cue exposure sessions, participants were asked to handle cocaine cues such as simulated crack, powder, and pipes while listening to an imagery script, and then they watched video footage of cocaine-related activities.
- DCS /DCS/Placebo: Participants were assigned to receive 50 mg of DCS at 2 cue exposure sessions, and placebo at the one-week follow-up session. During cue exposure sessions, participants were asked to handle cocaine cues such as simulated crack, powder, and pipes while listening to an imagery script, and then they watched video footage of cocaine-related activities. Cue exposure was accompanied by instructions on how to cope with craving.
- Placebo/Placebo/Placebo: Participants were assigned to receive placebo at 2 cue expsosure sessions, and at the one-week follow-up session. Participants also received cognitive skills training.During cue exposure sessions, participants were asked to handle cocaine cues such as simulated crack, powder, and pipes while listening to an imagery script, and then they watched video footage of cocaine-related activities. Cue exposure was accompanied by instructions on how to cope with craving.
- Total: Total of all reporting groups
Arm/Group | DCS/DCS/DCS/Placebo | Placebo/Placebo/Placebo/Placebo | DCS/ Placebo/DCS/Placebo | DCS /DCS/Placebo | Placebo/Placebo/Placebo | Total
Number analyzed (Participants) | 10 | 10 | 12 | 23 | 24 | 79
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 12 | 23 | 24 | 79
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.4 (10.9) | 45.1 (8.4) | 43.1 (5.9) | 49.1 (8.8) | 44.4 (8.7) | 45.5 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5 | 4 | 3 | 17
  Male | 9 | 6 | 7 | 19 | 21 | 62
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 12 | 23 | 24 | 79

OUTCOME MEASURES:

1. Primary Outcome: Subjective Craving of Cocaine
Description: Average of participants' subjective measures of craving immediately following cue exposure at the one-week follow-up session. Participants rated craving on a 10 point analog scale ranging from 0 (not at all) to 10 (extremely).
Time Frame: two weeks
Population: Data of participants who completed all cue exposure sessions and the one-week follow-up were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- DCS Only: Participants received 50 mg of DCS at each of 3 cue exposure sessions and placebo at the one-week follow-up session.
- Placebo Only: Participants received a placebo at each of 3 cue exposure sessions and at the one-week follow-up session.
- DCS/ Placebo/DCS: Participants received 50 mg of DCS at the 1st and 3rd cue exposure sessions, and placebo at the 2nd cue exposure session and the one-week follow-up session.
- DCS Plus Cognitive Skills Training: Participants received 50 mg of DCS at 2 cue extinction sessions and placebo at the one-week follow-up session. Participants also received cognitive skills training.
- Placebo Plus Cognitive Skills Training: Participants received a placebo at 2 cue extinction sessions and at the one-week follow-up session. Participants also received cognitive skills training.
Arm/Group | DCS Only | Placebo Only | DCS/ Placebo/DCS | DCS Plus Cognitive Skills Training | Placebo Plus Cognitive Skills Training
Number analyzed (Participants) | 10 | 10 | 12 | 23 | 24
units on a scale | 2.47 (2.39) | 0.90 (1.54) | 1.19 (1.58) | 1.06 (1.23) | 1.69 (2.24)

ADVERSE EVENTS:
Groups:
- DCS/DCS/DCS/Placebo: Participants were assigned to receive 50 mg of DCS for each of 3 cue exposure sessions and a placebo at the one-week follow-up session.
- Placebo/Placebo/Placebo/Placebo: Participants were assigned to receive a placebo for each of 3 cue exposure sessions and at the one-week follow-up session.
- DCS/ Placebo/DCS/Placebo: Participants were assigned to receive 50 mg of DCS at the 1st and 3rd cue sessions and placebo at the 2nd cue session and the one-week follow-up session.
- DCS /DCS/Placebo: Participants were assigned to receive 50 mg of DCS at 2 cue exposure sessions, and placebo at the one-week follow-up session.
- Placebo/Placebo/Placebo: Participants were assigned to receive placebo at 2 cue exposure sessions, and at the one-week follow-up session.
Arm/Group | DCS/DCS/DCS/Placebo | Placebo/Placebo/Placebo/Placebo | DCS/ Placebo/DCS/Placebo | DCS /DCS/Placebo | Placebo/Placebo/Placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/12 | 0/23 | 0/24
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/12 | 0/23 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No